CLINICAL TRIAL: NCT03064269
Title: CAR-T Therapy for Central Nervous System B-cell Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UnicarTherapy
Record Dates: First submitted 2017-02-18; First posted 2017-02-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: B-cell Acute Lymphocytic Leukemia
Keywords: CNS B cell acute lymphocytic leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): CD19 CAR-T cells treated central nervous system B-cell acute lymphocytic leukemia.
  Interventions: Biological: CD19 CAR-T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells — CNS leukemia is defined as unequivocal evidence of leukemic blasts in the cerebrospinal fluid by cytology or flow cytometry; cranial palsies or a nonhemorrhagic mass seen in cranial computed tomography or magnetic resonance imaging because of infiltration by leukemia cells

SUMMARY:
This study will evaluates the safety and efficacy of Chimeric antigen receptor T cells (CAR-T) in treating central nervous system B-cell acute lymphocytic leukemia.

DETAILED DESCRIPTION:
CNS leukemia is defined as unequivocal evidence of leukemic blasts in the cerebrospinal fluid by cytology or flow cytometry; cranial palsies or a nonhemorrhagic mass seen in cranial computed tomography or magnetic resonance imaging because of infiltration by leukemia cells

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19 positive central nervous system B-cell acute lymphocytic leukemia
2. ALT/ AST 《 3x normal
3. Creatinine 《 3x normal
4. Age:10-60.
5. Signed informed consent

Exclusion Criteria:

1. Active hepatitis B , hepatitis C or HIV infection
2. Uncontrolled active infection
3. Pregnancy or breast-feeding women
4. Survival less than four weeks

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete remission (CR) rate | Participants will be followed for the duration of the treatment, an expected average of 12 months
  The safety of the humanized CD19 CAR-T cells treatment will be evalated and the maximum tolerated dose will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen LY, Kang LQ, Zhou HX, Gao HQ, Zhu XF, Xu N, Yu L, Wu DP, Xue SL, Sun AN. Successful application of anti-CD19 CAR-T therapy with IL-6 knocking down to patients with central nervous system B-cell acute lymphocytic leukemia. Transl Oncol. 2020 Nov;13(11):100838. doi: 10.1016/j.tranon.2020.100838. Epub 2020 Jul 31. PMID 32745961